CLINICAL TRIAL: NCT04949061
Title: Culturally Adapted Cognitive Behavioral Intervention to Reduce Psychological Distress Among COVID-19 Survivors: A Randomized Controlled Trial
Brief Title: The Effectiveness of Culturally Adapted Cognitive Behavioral Intervention Among COVID-19 Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021.265.IRB1.091
Record Dates: First submitted 2021-07-01; First posted 2021-07-02 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2021-07

CONDITIONS: Psychological Distress; Quality of Life; Depressive Symptoms; Anxiety
Keywords: COVID-19; COVID-19 survivors; Psychological distress; Online intervention; Quality of life
MeSH Terms: conditions — Depression; Anxiety Disorders; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: Culturally Adapted Cognitive Behavioral Intervention (CA-CBI) (Experimental): The experimental group will receive an 8-session CA-CBI in an online group format.
  Interventions: Behavioral: Culturally Adapted Cognitive Behavioral Intervention (CA-CBI)
- Control Arm: Enhanced Treatment as Usual (ETA-U) (Other): The control group will receive the information about freely available psychological support options. Also, they will receive brief psychoeducation about the mental health problems and psychological distress via online leaflets. After all the measurements are completed, the control group will be able to receive the CA-CBI.
  Interventions: Other: Enhanced Treatment as Usual (ETA-U)

INTERVENTIONS:
Behavioral: Culturally Adapted Cognitive Behavioral Intervention (CA-CBI) — CA-CBI is an intervention based on Culturally Adapted Cognitive Behavioral Therapy (CA-CBT) which was developed by Devon Hinton. This trans-diagnostic intervention has a structured manual which can be culturally adapted and it will be used to decrease psychological distress and increase quality of life by targeting cognitive and behavioral changes.
  Arms: Intervention Arm: Culturally Adapted Cognitive Behavioral Intervention (CA-CBI)
Other: Enhanced Treatment as Usual (ETA-U) — Participants who receive ETAU will be provided a brief psychoeducation via online leaflets and will be informed about centers where they can receive free psychosocial support.
  Arms: Control Arm: Enhanced Treatment as Usual (ETA-U)

SUMMARY:
The effectiveness study for Culturally-Adapted Cognitive Behavioral Intervention (CA-CBI) will be conducted with individuals infected with and recovered from Coronavirus disease (COVID-19) to measure if this intervention is effective in decreasing the COVID-19 survivors' psychological distress. Potential participants will be given an informed consent and then, they will be included in a screening procedure to assess their eligibility. 86 participants (43 in experimental and 43 in control group-randomly assigned) who pass the screening procedure will be invited to the effectiveness study. The experimental group will receive an 8-session intervention while the control group will receive a brief psychoeducation about problems during COVID-19 pandemic and information about the freely available psychological support options. The measurements will be conducted three times; one week before, one week after and five weeks after the intervention.

DETAILED DESCRIPTION:
The COVID-19 pandemic has an enormous psychological impact worldwide. Individuals with suspected or confirmed COVID-19 have been defined as one of the most vulnerable groups suffering from psychological distress during the pandemic. Individuals who were infected with and recovered from COVID-19 had a significantly increased risk for developing psychiatric conditions such as anxiety and mood disorders, substance use disorders, and insomnia, even when comparing with individuals who had other respiratory tract infections. In addition, these psychiatric conditions remained elevated at the 6-month period for COVID-19 survivors. Therefore, COVID-19 survivors should be considered to be in need of an urgent intervention.

Considering the COVID-19 pandemic and future epidemics of other infectious diseases, more evidence-based psychosocial interventions should be implemented via online services. Group-based cognitive behavioral therapy (CBT) is one of the interventions identified as effective in decreasing adverse psychological outcomes of COVID-19 pandemic, as well as of Ebola and Severe acute respiratory syndrome (SARS). One of the forms of CBT is culturally adapted CBT (CA-CBT) developed by Hinton. CA-CBT is a trans-diagnostic method targeting cognitive and behavioral changes while emphasizing emotion regulation and psychological flexibility with some techniques such as mindfulness exercises, meditation, and applied stretching. In Turkey, CA-CBT was tested on adolescents and found to be effective in decreasing the adolescents' anxiety and depression symptoms.

The investigators propose to conduct a randomized controlled trial in order to implement culturally adapted cognitive behavioral intervention (CA-CBI) to COVID-19 survivors and evaluate the effectiveness of the intervention in reducing the psychological distress for this particular group. After the screening phase and baseline assessment, the investigators will randomly assign the eligible participants into two arms (CA-CBI and Enhanced Treatment as Usual) and deliver CA-CBI in an online group format to the experimental arm. The investigators will assess whether the psychological distress levels and common mental health problems of the COVID-19 survivors in the experimental arm are decreased compared to the control arm. The investigators will examine the study outcomes of the both arms at three times: Pre-assessment (1 week before the intervention), post-assessment (1 week after the intervention) and follow-up assessment (1 month after the post-assessment). A process evaluation according to the World Health Organization (WHO) will be completed with 5 study completers, 5 drop-outs and 2 facilitators to evaluate the feasibility of delivering CA-CBI.

To the knowledge, CA-CBI has not been conducted with survivors of an infectious disease before. Also, there are scarce publications on mental health interventions implemented to COVID-19 survivors. There is a need for more evidence-based psychological interventions that can be applied to the times of COVID-19 pandemic and future epidemics of infectious diseases, especially for vulnerable groups. Therefore, the investigators will contribute to the literature by applying online-delivered group-based CA-CBI to COVID-19 survivors with increased levels of psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or above
* Getting infected with COVID-19 and currently, recovered
* Scoring 16 or above on Kessler Psychological Distress Scale (K10)

Exclusion Criteria:

* Imminent suicidal risk
* Having a severe psychiatric disorder (psychotic disorders, acute mania, substance/alcohol addiction, cluster B personality disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Comparison of changes of the Kessler-10 Psychological Distress Scale (K10) over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)
  Kessler-10 Psychological Distress Scale is a 10-item scale that aims to measure the psychological distress. Each item is scored from 1 (none of the time) to 5 (all of the time) providing a range between 10 and 50. Higher scores indicate more severe psychological distress.

SECONDARY OUTCOMES:
Comparison of changes of the Patient Health Questionnaire-9 (PHQ-9) over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)
  Patient Health Questionnaire is a 9-item questionnaire that aims to measure the depressive symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day) providing a range between 0 and 27. Higher scores indicate more severe depressive symptoms.
Comparison of changes of the General Anxiety Disorder-7 (GAD-7) over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)
  General Anxiety Disorder-7 is a 7-item questionnaire that aims to measure anxiety symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day) providing a range between 0 and 21. Higher scores indicate higher levels of anxiety symptoms
Comparison of changes of the PTSD Checklist for The Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) (PCL-5) over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)
  The PTSD Checklist for DSM-5 is a 20-item questionnaire that assesses the symptoms of post-traumatic stress disorder. Each item is scored from 0 (not at all) to 4 (extremely) providing a range between 0 and 80. Higher scores indicate higher levels of PTSD symptoms.
Comparison of changes of the Symptom Checklist 90-R (SCL-90-R) Somatization Subscale over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)
  The SCL-90-R Somatization Subscale is a 12-item scale that measures somatic complaints based on self-report. Each item is scored from 0 (not at all) to 4 (extremely), providing a range between 0 and 48. Higher scores indicate higher levels of somatic complaints.
Comparison of changes of the World Health Organization Quality of Life Scale (WHOQOL Bref) over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)
  The WHOQOL Bref Scale is a 27-item questionnaire that assesses the quality of general health and life. It has four domains which are physical health, psychological health, social relationships, and environment. It also has questions about overall perceptions of life quality and general health. Each item is scored from 1 to 5 on a 5-point Likert scale. For each domain, the mean score is calculated, providing a range between 4 and 20. Each mean domain score is multiplied by 4 to transform the domain score into a scaled score. In each domain, higher scores indicate higher levels of quality of life.

OTHER OUTCOMES:
Comparison of changes of the Psychological Flexibility Scale over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)
  The Psychological Flexibility Scale is a 28-item scale that aims to assess psychological flexibility. Each item is scored from 1 (strongly disagree) to 7 (strongly agree), providing a range between 28 and 196. Higher scores indicate more frequent use of psychological flexibility in individuals.
Comparison of changes of the Emotion Regulation Questionnaire over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)
  The Emotion Regulation Questionnaire is a 10-item questionnaire that aims to measure individual differences in emotion regulation and its strategies. Each item is scored from 1 (strongly disagree) to 7 (strongly agree) providing a range between 10 and 70. It has two subscales which are re-appraisal and suppression. Higher scores indicate more frequent use of these strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Talya Öztürk, BA, Study Chair — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luo M, Guo L, Yu M, Jiang W, Wang H. The psychological and mental impact of coronavirus disease 2019 (COVID-19) on medical staff and general public - A systematic review and meta-analysis. Psychiatry Res. 2020 Sep;291:113190. doi: 10.1016/j.psychres.2020.113190. Epub 2020 Jun 7. PMID 32563745
- [Background] Acarturk ZC, Abuhamdeh S, Jalal B, Unaldi N, Alyanak B, Cetinkaya M, Gulen B, Hinton D. Culturally adapted transdiagnostic CBT for SSRI resistant Turkish adolescents: A pilot study. Am J Orthopsychiatry. 2019;89(2):222-227. doi: 10.1037/ort0000310. Epub 2018 Jan 18. PMID 29345479
- [Background] Kananian S, Soltani Y, Hinton D, Stangier U. Culturally Adapted Cognitive Behavioral Therapy Plus Problem Management (CA-CBT+) With Afghan Refugees: A Randomized Controlled Pilot Study. J Trauma Stress. 2020 Dec;33(6):928-938. doi: 10.1002/jts.22615. Epub 2020 Nov 5. PMID 33155348
- [Background] Hinton DE, Pham T, Tran M, Safren SA, Otto MW, Pollack MH. CBT for Vietnamese refugees with treatment-resistant PTSD and panic attacks: a pilot study. J Trauma Stress. 2004 Oct;17(5):429-33. doi: 10.1023/B:JOTS.0000048956.03529.fa. PMID 15633922
- [Background] Yue JL, Yan W, Sun YK, Yuan K, Su SZ, Han Y, Ravindran AV, Kosten T, Everall I, Davey CG, Bullmore E, Kawakami N, Barbui C, Thornicroft G, Lund C, Lin X, Liu L, Shi L, Shi J, Ran MS, Bao YP, Lu L. Mental health services for infectious disease outbreaks including COVID-19: a rapid systematic review. Psychol Med. 2020 Nov;50(15):2498-2513. doi: 10.1017/S0033291720003888. Epub 2020 Nov 5. PMID 33148347
- [Background] Taquet M, Geddes JR, Husain M, Luciano S, Harrison PJ. 6-month neurological and psychiatric outcomes in 236 379 survivors of COVID-19: a retrospective cohort study using electronic health records. Lancet Psychiatry. 2021 May;8(5):416-427. doi: 10.1016/S2215-0366(21)00084-5. Epub 2021 Apr 6. PMID 33836148
- [Background] Wang Y, Kala MP, Jafar TH. Factors associated with psychological distress during the coronavirus disease 2019 (COVID-19) pandemic on the predominantly general population: A systematic review and meta-analysis. PLoS One. 2020 Dec 28;15(12):e0244630. doi: 10.1371/journal.pone.0244630. eCollection 2020. PMID 33370404

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT04949061/Prot_SAP_002.pdf
  • Informed Consent Form (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT04949061/ICF_001.pdf